CLINICAL TRIAL: NCT01595399
Title: Atropine Versus no Atropine for Neonatal Rapid Sequence Intubation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R500458
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2012-05

CONDITIONS: Bradycardia; Hypoxemia
Keywords: bradycardia; hypoxemia; intubation; premedication
MeSH Terms: conditions — Bradycardia; Hypoxia | interventions — Atropine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Atropine, fentanyl and succinylcholine (Active Comparator): 20 mcg/kg atropine IV, 3 mcg/kg fentanyl slowly IV and 2 mg/kg succinylcholine IV.
  Interventions: Drug: atropine
- placebo, fentanyl and succinylcholine (Placebo Comparator): an equivalent volume of normal saline to atropine IV, 3 mcg/kg fentanyl slowly IV and 2 mg/kg succinylcholine IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atropine — Atropine 0.02 mg/kg IV
  Other Names: AtroPen
  Arms: Atropine, fentanyl and succinylcholine
Drug: Placebo — an equivalent volume of normal saline to atropine IV
  Other Names: 0.9% sodium chloride
  Arms: placebo, fentanyl and succinylcholine

SUMMARY:
The purpose of this study is to compare heart rate in infants who receive atropine as a part of their medication before intubation to those who do not.

To be able to find out , we need to divided babies into 2 groups;

group 1 : receives atropine + sedation + muscle relaxant group 2 : receives water or saline ( placebo group) + sedation + muscle relaxant

Then we need to compare heart rate during intubation and duration of intubation between the 2 groups.

DETAILED DESCRIPTION:
We hypothesize that premedication for intubation with fentanyl and succinylcholine alone will maintain equal stability of heart rate and oxygen saturation without a prolongation of time to completion of intubation when compared to a protocol using atropine, fentanyl and succinylcholine.

In order to answer this question we plan to undertake a prospective randomized double blinded control trial of use of atropine as an adjunct for elective intubation of infants less than 46 weeks postmenstrual age.

ELIGIBILITY:
Inclusion Criteria:

* Any infant (preterm and term) up to 46 weeks corrected age requiring (nonemergent) intubation.
* IV access is obtained
* Informed parental consent

Exclusion Criteria:

* Emergent intubation or need for resuscitation
* Congenital cyanotic heart disease
* Obvious airway abnormalities
* History of myopathy or family history of malignant hyperthermia or known history of phosphocholinesterase deficiency

Ages: 1 Day to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Heart rate less than 80 BPM and oxygen saturation less than 80% | 5-6 minutes
  Heart rate and transcutaneous oxygen saturation will be monitored continuously during the procedure and data will be recorded at 3 stages;
  1. 2 minutes prior to intubation (after atropine or placebo dose)
  2. during intubation
  3. 2 minutes after intubation (once ETT secured to face)

SECONDARY OUTCOMES:
Heart rate < 100 BPM | 5-6 minutes
Oxygen saturation < 85% | 5-6 minutes
Duration of intubation attempts | 1-2 minutes
Number of intubation attempts | 5-6 minutes
Lowest heart rate after premedication | 5-6 minutes
Lowest oxygen saturation after premedication | 5-6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Narvey, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Afifi J, El-Naggar W, Hatfield T, Sandila N, Baier J, Narvey M. Atropine Versus Placebo for Neonatal Nonemergent Intubation: A Randomized Clinical Trial. J Pediatr. 2025 Nov;286:114719. doi: 10.1016/j.jpeds.2025.114719. Epub 2025 Jul 9. PMID 40645282